CLINICAL TRIAL: NCT00568620
Title: The Role of the Duodenum in the Pathogenesis of Insulin Resistance and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Naji Abumrad, Chairman, Department of Surgery, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB#070770; R01DK070860 (NIH); GCRC #1710
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Insulin Resistance and Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Nasogastric feeding tube (Experimental)
  Interventions: Procedure: Placement of nasogastric feeding tube
- 2: Placement of nasojejunal feeding tube (Experimental)
  Interventions: Procedure: Nasojejunal feeding tube

INTERVENTIONS:
Procedure: Placement of nasogastric feeding tube — Glucose tolerance test via nasogastric feeding tube
  50 g glucose tolerance test on day 1; 50 g glucose tolerance test with 30 mL oil on day 2; Intravenous glucose tolerance test on day 3
  Arms: 1: Nasogastric feeding tube
Procedure: Nasojejunal feeding tube — Glucose tolerance test via nasojejunal feeding tube
  50 g glucose tolerance test on day 1; 50 g glucose tolerance test with 30 mL oil on day 2; Intravenous glucose tolerance test on day 3
  Arms: 2: Placement of nasojejunal feeding tube

SUMMARY:
In parallel with the increasing prevalence of obesity worldwide, type 2 diabetes mellitus (T2DM) has reached epidemic proportions. Despite a multitude of available therapies, only bariatric surgery (e.g., roux-en-Y gastric bypass (GBP)) has proven to be an effective long term treatment modality for morbid obesity. Moreover, the majority of T2DM patients who undergo GBP experience normalization of their blood glucose and are able to discontinue their anti-diabetes medications soon after the procedure. The insulin resistant state commonly seen in non-diabetic obese subjects also improves after GBP. Evidence from recent animal studies suggests that the rapid return to euglycemia seen in T2DM patients after GBP might in part result from excluding the duodenum from the flow of nutrients. With the use of enteral feeding tubes, we hope to better understand the factors in the human gut that may predispose obese individuals to the development of insulin resistance and T2DM.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for lean, healthy control subjects:

1. Fasting plasma glucose (FPG) < 100
2. Age 18 to 55
3. BMI 18.5 to 24.9 kg/m2
4. Stable weight for prior 3 months

Inclusion criteria for prediabetic individuals:

1. Based on American Diabetes Association criteria of FPG > 100 and <126
2. Age 18 to 55
3. BMI 35 to 60 kg/m2
4. Stable weight for prior 3 months

Inclusion criteria for diabetic individuals:

1. Diagnosis of type 2 diabetes mellitus (T2DM) for < 5 years
2. Hemoglobin A1c < 8%
3. Age 18 to 55
4. BMI 35 to 60 kg/m2
5. Stable weight for prior 3 months

Exclusion Criteria:

Exclusion criteria for all study subjects:

1. Use of any of the following medications: Thiazolidinediones, dipeptidyl-peptidase IV (DPP-IV) inhibitors (e.g., sitagliptin), GLP-1 analogs (e.g., exenatide).
2. Subjects with T2DM who are unable to maintain adequate glycemic control (i.e., having a fasting blood glucose that exceeds 250mg/dL on two consecutive tests) while temporarily discontinuing their oral diabetes medications for the study and in whom the study physician determines insulin therapy would not be appropriate.
3. Females with a positive pregnancy test

5. Prior gastric, duodenal, proximal jejunal surgery or pancreas resection 6. Known malabsorptive disorder 7. History of cancer in past 5 years 8. Renal insufficiency defined by serum creatinine > 1.5 mg/dl 9. Hepatic enzyme elevations of greater than twice the upper limits of normal 10. Current use of warfarin or clopidogrel 11. Intercurrent infections 12. Contraindication to nasogastric or nasojejunal feeding tube (e.g., deviated nasal septum, prior upper gastrointestinal bleed, or history of easy bleeding) 13. Residence outside the greater Nashville, TN area

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-05; Primary Completion 2012-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 3 days

SECONDARY OUTCOMES:
Incretin effect | 3 days

REFERENCES:
- [Derived] Tamboli RA, Sidani RM, Garcia AE, Antoun J, Isbell JM, Albaugh VL, Abumrad NN. Jejunal administration of glucose enhances acyl ghrelin suppression in obese humans. Am J Physiol Endocrinol Metab. 2016 Jul 1;311(1):E252-9. doi: 10.1152/ajpendo.00082.2016. Epub 2016 Jun 7. PMID 27279247